CLINICAL TRIAL: NCT02565433
Title: Prospective Assessment of Quality of Life in Patients Treated by Radiosurgery for Brain Metastases
Brief Title: Prospective Assessment of Quality of Life in Patients Treated by Radiosurgery for Brain Metastases (PRAMECE-1302)
Acronym: PRAMECE-1302
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PRAMECE-1302
Record Dates: First submitted 2015-05-19; First posted 2015-10-01 (Estimated); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Neoplasm Metastases
Keywords: brain metastases; Gamma Knife; Radiosurgery; Quality of Life
MeSH Terms: conditions — Neoplasm Metastasis; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- questionnaire administration (Experimental): Quality of life questionnaires administration (EORTC QLQ C30 and BN20 / IADL / HADS / MoCa Edmonton Symptom Assessment Scale)
  Interventions: Other: questionnaire administration

INTERVENTIONS:
Other: questionnaire administration — Within 15 days before radiosurgery and then at 3, 6, 9, 12 months after radiosurgery, the patients who have accepted to participate will have to complete these questionnaires : QLQC30, BN20, IADL, HADS, MoCa, Edmonton Symptom Assessment Scale
  Other Names: survey administration

SUMMARY:
The aim of the study is to assess prospectively the impact of radiosurgery on the quality of life in patients with brain metastases.

DETAILED DESCRIPTION:
The patients who meet the selection criteria and who have accepted to participate at the study will answer different questionnaires of the study before radiosurgery and at 3, 6, 9 and 12 months after the treatment of brain metastases. Baseline examinations will be done before receiving the treatment during the hospitalisation for the Gamma Knife treatment, and then they will be repeated at the evaluation visits which are classically done every 3 months. MRI's will also be performed every 3 months. In this way, no additional travel or MRI will be carried out as part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient with newly diagnosed brain metastases
* Patient with cancer regardless of the type of primary cancer, with anatomopathological proof
* At least, one measurable lesion ≥ 10 mm on the MRI T1 gadolinium sequences
* Number of brain metastases lower or equal to 5
* Indication of radiosurgery treatment
* Age ≥ 18 years old
* ECOG-PS 0-2
* Expected survival > 3 months
* Ability to complete self-administered questionnaires. If the patient has a motor disability (hemibody deficit) that does not allow to complete himself the questionnaires, these will be read by a CRA of the Neurosurgery department who will outline the questions without making any comment.
* A non-opposition form must have been completed by the patient

Exclusion Criteria:

* Previous cancer (< 5 years) except of carcinoma of cervix uteri, basal cell or squamous cell skin carcinoma adequately treated
* Previous brain radiotherapy
* Neurological pathology with cognitive disorders existing before the study
* Having a contraindication for MRI
* Associated leptomeningeal disease
* Patients having another severe or uncontrolled pathology which could compromise the participation at the study (such as infection, cardiovascular, digestive, renal or pulmonary disease)
* Pregnant or breastfeeding woman. The women must not breastfeed for at least 6 months
* Impossibility to submit to the medical examinations of the study due to geographic, social or mental reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-11; Primary Completion 2018-01 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Impact at 6 months of the radiosurgery based on the evaluation of 4 criteria of the QLQ C30 questionnaire | 6 months
  The 4 criteria are the perceived overall state, health, physical functioning, cognitive functioning and tiredness

SECONDARY OUTCOMES:
Comparison of the scores obtained on the scales, questionnaires and Performance status at baseline and every 3 months (until 12 months) after Gamma Knife treatment | 1 year
  QLQ C30, BN20 (quality of life), IADL (autonomy), HADS (anxiety-depression), MoCA (cognition), ESAS (quality of life), Performance status (OMS)
Comparison of the scores obtained on the scales and questionnaires according to the type of primary cancer at baseline and every 3 months (until 12 months) after Gamma Knife treatment | 1 year
  QLQ C30, BN20 (quality of life), IADL (autonomy), HADS (anxiety-depression), MoCA (cognition)
Comparison of the scores obtained on different scales according to the type of associated treatments at baseline and every 3 months (until 12 months) after Gamma Knife treatment | 1 year
  The type of associated treatments are: chemotherapy, targeted therapy, corticoids, anti-epileptics, psychotropic drugs.
  The different scales are QLQ C30, BN20 (quality of life), IADL (autonomy), HADS (anxiety-depression), ESAS (quality of life) and MoCA (cognition)
Correlation between the scores obtained on the different scales at the baseline and the progression-free survival / overall survival | 1 year
Correlation between the scores obtained on the scales QLQ C30, BN20 (quality of life), IADL (autonomy), HADS (anxiety-depression), MoCA (cognition), ESAS (quality of life) at baseline and those obtained at 3, 6, 9, 12 months | 1 year
Correlation between the scores obtained on the scales during the study and the clinical neurological response at baseline and every 3 monts until 12 months after Gamma Knife treatment | 1 year
  The correlation will take into account the evolution of the systemic disease and the volumetric tumor response. Volumetric tumor responses will be calculated on the MRI's

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Le Rhun, MD, Principal Investigator — Centre Oscar Lambret; Franck Bonnetain, MD, Study Director — CHRU de Besançon
Locations (1):
- CHRU de Lille - Hôpital Salengro, Lille, France

IPD SHARING:
Plan to Share IPD: No